CLINICAL TRIAL: NCT06892301
Title: Clinical Exploration Study of YOLT-203 in the Treatment of Type 1 Primary Hyperoxaluria (PH1)
Acronym: PH1
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH1-YOLT-203-01
Record Dates: First submitted 2025-02-26; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Primary Hyperoxaluria
MeSH Terms: conditions — Primary hyperoxaluria type 1

STUDY DESIGN:
Intervention Model Description: 0.45mg/kg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label single dose (Experimental): YOLT-203
  Interventions: Drug: YOLT-203

INTERVENTIONS:
Drug: YOLT-203 — The IP is administered intravenously at the predetermined dose.

SUMMARY:
This study is a single-arm, open-label, single-dose, dose-escalation trial, aiming to evaluate the safety and tolerability of YOLT-203 in the Chinese population with type 1 primary hyperoxaluria (PH1); and to preliminarily assess the effect of a single dose of YOLT-203 on the plasma oxalate level.In this study, the maximum screening period of the main study is 60 days, the treatment day is Day 1 (D1), and the safety follow-up period is up to Week 52 after administration. In addition, subjects within the first dose group can voluntarily receive a second treatment with the test drug at the effective dose level. After the end of the main study, the subjects will undergo long-term followup. According to the requirements of the "Technical Guidelines for Long-Term Follow-up Clinical Studies of Gene Therapy Products (Trial)" issued by the CDE, the long-term follow-up is up to 15 years after administration. The most updated protocol is V1.2 , 22 Jan 2025

ELIGIBILITY:
Inclusion Criteria:

* The age is 2≤ years <18 years old at the time of signing the informed consent.

  * Have AGXT gene mutations and be diagnosed with primary hyperoxaluria (PH1); eGFR ≥ 30 ml/min/1.73m2.
  * At least 2 times of 24-hour urinary oxalate excretion ≥ 0.7 mmol/1.73m2/ day or the ratio of urinary oxalate to creatinine in a single urine collection must be higher than the upper limit of normal (ULN) for the corresponding age.
  * If treated with vitamin B6, the treatment has been stable for 90 days before enrollment in the study and is willing to maintain the stable treatment plan unchanged during the study.
  * The patient himself/herself or the guardian voluntarily signs the informed consent.

Exclusion Criteria:

* The investigator judges that there is clinical evidence of systemic extrarenal oxalate deposition.

  * Have any of the following laboratory parameter assessment results at screening:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x the upper limit of normal (ULN).
    2. Total bilirubin > 1.5 x ULN. If the increase in total bilirubin is caused by diagnosed Gilbert's syndrome and the total bilirubin < 2 x ULN, it is eligible.
    3. International normalized ratio (INR) > 1.5 (Patients on oral anticoagulants [such as warfarin] and with INR < 3.5 will be allowed to participate).
  * Known to have active human immunodeficiency virus (HIV) infection; or have evidence of current or chronic hepatitis C virus (HCV) or hepatitis B virus (HBV) infection.
  * The estimated glomerular filtration rate (GFR) at screening is less than 30 mL/min/1.73m² (For patients ≥ 18 years old, it will be calculated according to the Modification of Diet in Renal Disease [MDRD] formula; for patients < 18 years old, it will be calculated according to the Schwartz bedside formula). See the attachment.
  * Have received an investigational drug within the last 30 days or 5 halflives (whichever is longer) before the first administration of the study drug, or have participated in the follow-up of another clinical study before randomization.
  * Have a history of kidney or liver transplantation.
  * According to the investigator's opinion, have other medical conditions or comorbidities that may interfere with study compliance or data interpretation.
* Page 4 of 5 [DRAFT] -

  * Have a history of multiple drug allergies or allergic reaction history to oligonucleotides or LNP.
  * Have a history of subcutaneous injection intolerance.
  * Unwilling to comply with contraceptive requirements throughout the study participation period until 6 months after the end of the main study trial.
  * Female patients are pregnant, planning to become pregnant or breastfeeding.
  * Unwilling or unable to limit alcohol consumption throughout the study. Alcohol consumption during the study exceeds 2 units per day (1 unit: approximately 125 ml of wine = approximately 29 ml of spirits = approximately 284 ml of beer, will be excluded.
  * The investigator believes that there is a history of alcohol abuse within 12 months before screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse events | through week 52
  An Adverse Event(AE) is any untoward medical occurrence in a participant or clinical investigational participant adminstered a medicinal product and which does not necessarily have a casual relationship with this treatment

SECONDARY OUTCOMES:
The Peak Plasma Concentration (Cmax) of YOLT-203 | through Day 14
  The Peak Plasma Concentration (Cmax) of YOLT-203 in the plasma after a dose is given
Area under the plasma concentration versus time curve (AUC)of YOLT-203 | through Day 14
  Area under the plasma concentration versus time curve (AUC). 0.5 predose,6,24,48,144,and312 hours after treatment
Time to Maximum Plasma Concentration (Tmax)of YOLT-203 | through Day 14
  Tmax is the time it takes for YOLT-203 to reach the maximun concentration (Tmax) after administration
Drug half-life (T1/2)of YOLT-203 | through Day 14
  The amount of time it takes for the plasma YOLT-203 drug concentration to drop to half
The changes in blood glycolic acid levels | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in blood glycolic acid levels
The changes in 24-hour urinary oxalic acid excretion | through week 52
  After medication, at 1,2,4, 8, 16, 24, 36and 52 weeks, the changes in 24-hour urinary oxalic acid excretion compared to the baseline value.
The changes in 24-hour urinary glycolic acid excretion | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in 24-hour urinary glycolic acid excretion
The changes in eGFR | through week 52
  After medication, at 1, 2, 4, 8, 16, 24, 36, and 52 weeks, the changes in eGFR.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, PhD, MD, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China